CLINICAL TRIAL: NCT03745378
Title: Secondary Cancers in Myeloproliferative Neoplasms (MPN-K Study)
Acronym: MPN-K
Status: Completed | Type: Observational
Sponsor: FROM- Fondazione per la Ricerca Ospedale di Bergamo- ETS (Other)
Responsible Party: Sponsor
Other Study IDs: MPN-K - FROM/O2- 2017
Record Dates: First submitted 2018-10-15; First posted 2018-11-19 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Polycythemia Vera; Essential Thrombocythemia; Myelofibrosis
Keywords: Myeloproliferative neoplasms; Secondary cancer; JAK2V617F mutation
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential; Primary Myelofibrosis; Myeloproliferative Disorders; Neoplasms, Second Primary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients with diagnosis of Myeloproliferative Neoplasms (MPN) including Polycythemia Vera, Essential thrombocytopenia or Myelofibrosis, exposed or not exposed to JAK2V617F mutation, who experienced secondary cancer(s) diagnosed at presentation of MPN or during the course of the myeloproliferative disease.
  Interventions: Other: JAK2V617F mutation
- Controls: Patients with diagnosis of Myeloproliferative Neoplasms (MPN) including Polycythemia Vera, Essential thrombocytopenia or Myelofibrosis, exposed or not exposed to JAK2V617F mutation, without history of secondary cancer.
  Interventions: Other: JAK2V617F mutation

INTERVENTIONS:
Other: JAK2V617F mutation — JAK2 V617F is attached to the cytosolic juxtamembrane region of dimeric cytokine receptors, such as EpoR or MPL (TpoR); The JAK2V617F mutation results from a guanine to thymine change at nucleotide 1849 of the cDNA, in exon 14 of the gene. This valine is located at one of the predicted interfaces between JH1 and JH2 domains,

SUMMARY:
The incidence of secondary cancer (SC) in patients with myeloproliferative neoplasms (MPN) is high and comparable to that of thrombosis. However, the identification of patient subgroups that might be at increased susceptibility of developing SC has not been systematically addressed. This international case-control study (MPN-K) is aimed to elucidate the prognostic role of JAK2V617F mutation in predicting the occurrence of SC in patients with classical MPN, polycythemia vera (PV), essential thrombocythemia (ET) and myelofibrosis (MF)

DETAILED DESCRIPTION:
For each recruited case with concomitant diagnosis of myeloproliferative neoplasms (MPN) and secondary cancer each participating center will provide up 3 control patients (1 control for each case could be accepted but the optimal number is 3). Controls are patients with myeloproliferative neoplasms and no history of cancer. Each control will be matched to the paired case for sex, age (+/- 3 years), date of MPN diagnosis (+/- 5 years), and MPN disease duration (+/- 3 years).

Each control is censored at the date of the secondary cancer occurrence in his matched case (index date).

Data will be collected retrospectively from pre-existing medical records and reported by each center on a web-based and validated eCRF developed to record y all study data. In order to maintain patient privacy, all data records will be treated anonymously and no personal data to identify patient will be recorded: patients will be identified in the study by an alphanumeric code.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Philadelphia-negative Myeloproliferative Neoplasms (MPN) according to PVSG, 2008 and 2016 WHO criteria, including:
* Polycythemia Vera (PV)
* Essential Thrombocythemia (ET)
* Myelofibrosis (MF), including both primary and secondary MF
* Diagnosis performed between 1st January 2000 to 31 December 2016
* Diagnosis of secondary cancer(s) performed concurrently or subsequently the diagnosis of MPN

Exclusion Criteria:

- Diagnosis of cancer occurred before the diagnosis of MPN (PV, ET, MF)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Matching characteristics for inclusion: sex, age at diagnosis of MPN (+/-3 years), date of MPN diagnosis (+/- 5 years), and MPN disease duration (+/- 3 years).
Sampling Method: Non-Probability Sample
Enrollment: 1881 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2018-07-07 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with secondary cancers after diagnosis of Polycythemia Vera (PV), Essential Trombocythemia (ET) and Myelofibrosis (MF) | 10 year from diagnosis of PV, ET or MF
  The ratio of number of patients showing JAK2V617F mutation on the number of patients not exposed to this mutation will be calculated in the group of subjects experiencing second cancer after diagnosis of PV, ET and MF (defined as 'cases') and related (odds ratio) with the ratio of patients exposed on those not exposed to JAK2V617F mutation in the group of subjects with no experience of secondary cancers after diagnosis of PV, ET and MF (this group is defined as 'Control' group)

SECONDARY OUTCOMES:
Number of patients with secondary cancers after diagnosis of Polycythemia Vera (PV), Essential Trombocythemia (ET) and Myelofibrosis (MF) in subgroups of subjects exposed to potential risk factors at diagnosis | 10 year from diagnosis of PV, ET or MF
  Characteristics at diagnosis of patients with PV, ET and MF (including other mutations) with occurrence of second cancers (SC) are decribed and compared with those not experiencing SC after diagnosis of myloproliferative neoplasm; the ratio of number of patients exposed to potential risk factors on the number of subjects not exposed will be calculated in the group cases (as defined for primary outcome measure) and related (odds ratio) with the ratio of patient exposed versus not exposed calculated in the subgroup of control.
Number of patients with secondary cancers after diagnosis of Polycythemia Vera (PV), Essential Trombocythemia (ET) and Myelofibrosis (MF) in the subgroups exposed to treatment | 10 year from diagnosis of PV, ET or MF
  Group of patients exposed and not exposed to different class of treatments for PV, ET and MF are compared and related in the group of cases and control

CONTACTS AND LOCATIONS:
Overall Officials: Tiziano Barbui, Prof, Study Chair — FROM- Fondazione per la Ricerca Ospedale di Bergamo- ETS; Guido Finazzi, Dr, Principal Investigator — ASST-Papa Giovanni XXIII
Locations (30):
- Palacky University and University Hospital Olomouc, Faculty of Medecine, Olomouc, Czechia
- Germany (2):
  - University Hospital RWTH - Department Oncology, Hematology, Hemostaeseology and stem cell transplantation, Aachen
  - Johannes Wesling Academic Medical Center, Minden
- Meir Medical Center, Kfar Saba, Israel
- Italy (18):
  - Azienda Sanitaria di Asti - A.S.L. AT Ospedale Cardinal Massaia - S.C. Oncologia, Asti
  - ASST- Papa Giovanni XXIII - UOC Ematologia, Bergamo
  - Ospedale S. Orsola - Malpighi - UO Ematologia, Bologna
  - U.O. Emostasi "G. Rodolico" Dipartimento di Scienze Mediche, Chirurgiche e Tecnologiche Avanzate "G.F. Ingrassia" Università degli Studi di Catania, Catania
  - Azienda Ospedaliera S. Croce e Carle di Cuneo- Divisione di Ematologia,, Cuneo
  - AOU Careggi di Firenze CRIMM- Center of Research and Innovation of Myeloproliferative Neoplasms - Department of Experimental and Clinical Medicine, University of Florence, Florence
  - Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico - UOC Ematologia, Milan
  - IRCCS Ospedale San Raffaele Unità Operativa di Ematologia e Trapianto Midollo Osseo, Milan
  - ASST MONZA Ospedale San Gerardo Clinica Ematologica, Monza
  - Azienda Ospedaliera Universitaria Federico II di Napoli Divisione di Ematologia e Trapianti del Midollo, Napoli
  - Azienda Ospedaliero Universitaria Maggiore della Carità di Novara SCDU Ematologia, Novara
  - Fondazione IRCCS Policlinico San Matteo S.C Ematologia, Pavia
  - AUSL IRCCS di Reggio Emilia Presidio Osp. Arcispedale Santa Maria Nuova - Unità Ematologia, Reggio Emilia
  - Fondazione Policlinico Universitario A. Gemelli IRCCS UCSC Ematologia, Roma
  - A.O.U. Città della Salute e della Scienza di Torino - Ospedale Molinette- S.C. Ematologia, Torino
  - A.O.U. Città della Salute e della Scienza di Torino Ospedale Molinette - S.C. Ematologia U, Torino
  - Ospedale Borgo Roma - Unità di Ematologia, Verona
  - Ospedale San Bortolo di Vicenza - U.O.C di Ematologia, Vicenza
- Spain (6):
  - Hospital Clinic, Hematology Department, Barcelona
  - Hospital del Mar - Haematologia Clinica, Barcelona
  - Hospital Universitario Vall d' Hebron - Unit Hematology, Barcelona
  - University Clinical Hospital of Santiago De Campostela - Service of Hematology, Santiago de Compostela
  - Hospita Clinico Universitario - Hematology Department, Valencia
  - Miguel Servet University Hospital, Zaragoza
- United Kingdom (2):
  - Belfast Health and Social Care Trust - Unit Haematology, Belfast
  - Guy's and St Thomas' NHS Foundation Trust, London

REFERENCES:
- [Derived] De Stefano V, Ghirardi A, Masciulli A, Carobbio A, Palandri F, Vianelli N, Rossi E, Betti S, Di Veroli A, Iurlo A, Cattaneo D, Finazzi G, Bonifacio M, Scaffidi L, Patriarca A, Rumi E, Casetti IC, Stephenson C, Guglielmelli P, Elli EM, Palova M, Rapezzi D, Erez D, Gomez M, Wille K, Perez-Encinas M, Lunghi F, Angona A, Fox ML, Beggiato E, Benevolo G, Carli G, Cacciola R, McMullin MF, Tieghi A, Recasens V, Isfort S, Marchetti M, Griesshammer M, Alvarez-Larran A, Vannucchi AM, Rambaldi A, Barbui T. Arterial thrombosis in Philadelphia-negative myeloproliferative neoplasms predicts second cancer: a case-control study. Blood. 2020 Jan 30;135(5):381-386. doi: 10.1182/blood.2019002614. PMID 31869407